CLINICAL TRIAL: NCT04310241
Title: Oculomotor Disorders: Experimental and Clinical Study
Brief Title: Visual Function Abnormalities in Strabismus and Amblyopia and Response to Therapy
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Fatema Ghasia, Associate Staff, The Cleveland Clinic
Other Study IDs: 12-915
Record Dates: First submitted 2020-03-11; First posted 2020-03-17 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Amblyopia; Strabismus
MeSH Terms: conditions — Amblyopia; Strabismus | interventions — Eyeglasses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control subjects: Subjects who state they have no eye or neurologic problems or disease other than perhaps wearing glasses or contact lenses and upon review of medical history.
- Amblyopia: Clinical diagnosis of amblyopia
  Interventions: Behavioral: Patching therapy, Glasses

INTERVENTIONS:
Behavioral: Patching therapy, Glasses — Patching, glasses and strabismus surgery are commonly employed measures in treatment of amblyopia and strabismus.
  Other Names: Strabismus surgery
  Groups: Amblyopia

SUMMARY:
Amblyopia and strabismus are characterized by a reduction in visual acuity, contrast sensitivity, grating acuity, vernier acuity, reading difficulties and binocular visual function deficits. Treated patients have residual visual function deficits. The purpose of the current study is to quantify various visual functions in amblyopic and strabismic participants at baseline, during and at the completion of treatment.

DETAILED DESCRIPTION:
To examine the response of therapy on visual functions in amblyopic and strabismic participants.

The following visual functions will be measured prior to treatment. Eye movements, contrast sensitivity, grating acuity, visual acuity, vernier acuity, binocular visual functions, reading and visual scanning will be measured. The testing will comprise of one or more of the above paradigms depending on participant's cooperation and understanding as majority of the study participants will be children. The above measurements will be repeated during amblyopia therapy ( which comprises of glasses, patching and/or atropine eye drops) and at the completion of treatment. For participants with strabismus requiring strabismus surgery the measurements will be repeated after strabismus surgery.

ELIGIBILITY:
Inclusion Criteria:

* History of amblyopia or presence of amblyogenic risk factors.

Exclusion Criteria:

* History of neurologic disorders

Ages: 6 Months to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children with diagnosis of strabismus and/or amblyopia
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-02-21 (Actual); Primary Completion 2027-03-12 (Estimated); Study Completion 2027-03-12 (Estimated)

PRIMARY OUTCOMES:
Visual Functions | 0-3 years depending on duration of treatment
  contrast sensitivity
Visual Functions | 0-3 years depending on duration of treatment
  visual acuity
Visual functions | 0-3 years depending on duration of treatment
  vernier acuity
Visual functions | 0-3 years depending on duration of treatment
  grating acuity
Visual functions | 0-3 years depending on duration of treatment
  binocular functions- stereopsis, inter-ocular functions
Visual functions | 0-3 years depending on duration of treatment
  eye movement measurements
Visual functions | 0-3 years depending on duration of treatment
  reading- reading speeds, eye movement measurements

CONTACTS AND LOCATIONS:
Overall Officials: Fatema Ghasia, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Research publications require inclusion of de-identified data in the manuscript. We will also be presenting the data at local, national and international conferences.
Supporting Information: SAP, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: The de-identified research data will be shared with colleagues and will be published after peer-review.

REFERENCES:
- [Background] Shaikh AG, Otero-Millan J, Kumar P, Ghasia FF. Abnormal Fixational Eye Movements in Amblyopia. PLoS One. 2016 Mar 1;11(3):e0149953. doi: 10.1371/journal.pone.0149953. eCollection 2016. PMID 26930079
- [Background] Ghasia FF, Otero-Millan J, Shaikh AG. Abnormal fixational eye movements in strabismus. Br J Ophthalmol. 2018 Feb;102(2):253-259. doi: 10.1136/bjophthalmol-2017-310346. Epub 2017 Jul 11. PMID 28698242
- [Background] Chatzistefanou KI, Theodossiadis GP, Damanakis AG, Ladas ID, Moschos MN, Chimonidou E. Contrast sensitivity in amblyopia: the fellow eye of untreated and successfully treated amblyopes. J AAPOS. 2005 Oct;9(5):468-74. doi: 10.1016/j.jaapos.2005.05.002. PMID 16213398